CLINICAL TRIAL: NCT03587740
Title: ATOP TRIAL: Adjuvant Ado-Trastuzumab Emtansine (T-DM1) for Older Patients With Human Epidermal Growth Factor Receptor 2 (HER2)-Positive Breast Cancer
Brief Title: ATOP TRIAL: T-DM1 in HER2 Positive Breast Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Susan G. Komen Breast Cancer Foundation (Other); Gateway for Cancer Research (Other)
Responsible Party: Principal Investigator, Rachel Freedman, MD, MPH, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18-124; NCT02414646 (obsolete NCT alias)
Record Dates: First submitted 2018-06-21; First posted 2018-07-16 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Breast Cancer
Keywords: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Ado-Trastuzumab Emtansine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- T-DM1 (Experimental): T-DM1 will be administered every 3 weeks intravenously, with 21 consecutive days defined as a treatment.
  Interventions: Drug: T-DM1

INTERVENTIONS:
Drug: T-DM1 — T-DM1 is an antibody-drug conjugate; it is made up of an antibody (trastuzumab) linked to a cytotoxic drug, DM1 (chemotherapy). T-DM1 functions as a targeted cancer therapy because it targets HER2-positive breast cancer cells directly, limiting exposure of the rest of the body to chemotherapy.
  Other Names: Kadcyla

SUMMARY:
This research study is studying an investigational drug as a possible treatment for breast cancer that is positive for the protein Human Epidermal Growth Factor Receptor 2, also known as HER2-positive breast cancer.

The drug involved in this study is:

-ado-trastuzumab emtansine (T-DM1)

DETAILED DESCRIPTION:
This research study is a Phase II clinical trial. Phase II clinical trials test the safety and effectiveness of an investigational drug to learn whether the drug works in treating a specific disease. "Investigational" means that the drug is being studied and research doctors are trying to find out more about it-such as the safest dose to use and the side effects it may cause.

The purpose of this research study is to examine the long-term benefits of T-DM1 with regard to breast cancer and take a closer look at the side effects experienced by participants receiving T-DM1.

The FDA (the U.S. Food and Drug Administration) has not approved T-DM1 for use in patients with stage I, II, or III breast cancer, but it has been approved for use in advanced, previously treated, HER2-positive breast cancer.

T-DM1 is an antibody-drug conjugate; it is made up of an antibody (trastuzumab) linked to a cytotoxic drug, DM1 (chemotherapy). T-DM1 functions as a targeted cancer therapy because it targets HER2-positive breast cancer cells directly, limiting exposure of the rest of the body to chemotherapy. More specifically, the trastuzumab in T-DM1 first binds to the HER2 protein on the surface of the breast cancer cells and the DM1 then enters the cells and can cause them to die, preventing tumor growth

ELIGIBILITY:
Inclusion Criteria:

* Participants must have histologically or cytologically confirmed HER2-positive disease by local pathology, defined as immunohistochemistry (IHC) 3+ or amplification by FISH (HER2/CEP17 ratio ≥2 or an average of ≥6 HER2 gene copies per nucleus) AND confirmed by Central Pathology Review (Dr. Deborah Dillon at Brigham and Women's Hospital, Boston, MA) prior to patient being registered to begin protocol therapy. See section 3.4. http://ascopubs.org/doi/full/10.1200/jco.2013.50.9984
* NOTE: DCIS components should not be counted in the determination of HER2 status.
* Age ≥60 years at the time of study registration (men and women eligible)
* Participants must have histologically or cytologically confirmed Stage I-III breast cancer with the following criteria met:
* If node-negative or if node status unknown (because it was not assessed), tumor must be >5 mm of any hormone receptor subtype (document ER/PR status: if some ER/PR staining is present, ER and PR negative are defined as being positive in <10% cells [per local pathology read]).
* If node-positive (N1-N3), T1mi, T1a, T1b, T1c, T2, or T3 tumors are eligible (see below for further details on defining node-negative disease) Definition of node-negative disease (when node status known): If the patient has had a negative sentinel node biopsy and/or a negative axillary dissection, then the patient is determined to be node-negative. Axillary nodes with single cells or tumor clusters ≤ 0.2 mm by either H&E or IHC will be considered node-negative. Any axillary lymph node with tumor clusters between 0.02 and 0.2cm is considered a micrometastasis. Patients with a micrometastasis are eligible even if their tumor is </= 5mm. An axillary dissection is not required to be performed in patients with a positive sentinel node and management of the axilla will be left up to the treating provider. In cases where the specific pathologic size of lymph node involvement is subject to interpretation, the principal investigator will make the final determination as to eligibility. In these special situations, the investigator must document this approval in the patient medical record.
* ER/PR determination assays performed by IHC methods according to the local institution standard protocol.
* Standard chemotherapy/trastuzumab declined by patient OR patient is deemed by physician for any reason to not be a candidate for standard therapy (i.e. patient and/or provider choose not to pursue standard trastuzumab-based chemotherapy regimen because of concerns related to toxicity or provider/patient preference).
* For patients with bilateral or multifocal/multicentric breast cancers, one of the following criteria must be met to enroll: (1) each cancer individually meets criteria for enrollment (only ONE tumor has to undergo central confirmation for HER2), (2) at least one tumor meets eligibility (per tumor size/nodes/subtype outlined above) and the other foci in the ipsilateral or contralateral breast are also HER2-positive but are too small for enrollment (e.g., a patient is eligible if a cancer is T2N0 and HER2-positive in one breast, but the contralateral breast has a T1a HER2+ cancer that isn't eligible on its own, (3) there is at least one qualifying tumor of >5mm but there are other small foci of disease that are too small to test for ER/PR/HER2 and are felt to be a part of the same tumor or similar tumor, OR (4) at least one tumor meets eligibility and the other foci in the ipsilateral or contralateral breast are HER2-negative and do not meet criteria for adjuvant chemotherapy per provider discretion (e.g. if a patient has a HER2-positive tumor meeting eligibility but also has a second, HER2-negative, small, node-negative, ER+, low grade cancer present, she is still eligible for enrollment). However, in the specific case that a second breast cancer is stage III and HER2-negative, that patient is excluded (because the second cancer is high-risk and likely will require non-HER2-directed therapy).
* All tumor removed by either a modified radical mastectomy or a segmental mastectomy (lumpectomy).
* NOTE: Management of axillary lymph nodes is up to the treating provider; however, all surgical margins should be clear of invasive cancer or DCIS (i.e., no tumor on ink). The local pathologist must document negative margins of resection in the pathology report. If all other margins are clear, a positive posterior (deep) margin is permitted, provided the surgeon documents that the excision was performed down to the pectoral fascia and all tumor has been removed. Likewise, if all other margins are clear, a positive anterior (superficial; abutting skin) margin is permitted provided the surgeon documents that all tumor has been removed.

  -≤90 days from the patient's most recent breast surgery for this breast cancer. Note: In cases where registration will occur >90 days from surgery but within an acceptable time frame, patient may be eligible for enrollment with approval from the PI, Rachel Freedman MD, MPH.
* ECOG Performance Status (PS) 0-2. See Appendix F.
* Baseline ejection fraction ≥50% by MUGA scan or echocardiogram performed ≤60 days prior to registration.
* The following laboratory values obtained ≤14 days prior to registration:

  * Absolute neutrophil count (ANC) ≥1500/mm3
  * Platelet count ≥100,000/mm3
  * Hemoglobin >9.0 g/dL
  * Total bilirubin ≤1.5 x upper limit of normal (ULN). If patient has known Gilbert's syndrome, the suggested threshold for treatment is a total bilirubin ≤2.0 x ULN, but will be left to the treating providers discretion.
  * AST and ALT ≤2.5 x ULN, alkaline phosphatase ≤2.5 x ULN
  * INR <1.5 x ULN for institution unless patient is on planned therapy with anticoagulants (i.e., warfarin) with higher target planned. In those cases, INR up to 3.5 is acceptable.
  * PTT <1.5 x ULN for institution unless patient is on planned therapy with heparin or heparin-like products Note: In the case of longstanding ethnic neutropenia, patient may be eligible for enrollment with approval from the PI, Rachel Freedman MD, MPH.
* Life expectancy >5 years per provider's assessment
* Willing to employ adequate and appropriate birth control if applicable
* NOTE: This study is for patients aged 60 and older, and most female patients will have entered menopause by this time; however patients should not become pregnant while on this study because T-DM1 can affect an unborn baby. Pre-menopausal women need to use birth control while on this study and women should not breastfeed a baby while on this study. Any man treated on this study will also need to use contraception if his partner is a premenopausal female. Patients should check with their health care provider about what kind of birth control methods to use and how long to use them.
* Negative urine or serum pregnancy test done ≤7 days prior to registration, for women of childbearing potential only
* NOTE: In the rare case that a woman enrolling on study is of childbearing potential, a pregnancy test is required prior to enrollment on study.
* Able to provide informed written consent.
* Willing to return to consenting institution for follow-up at 6 months
* Willing to provide blood samples for mandatory correlative research purposes.
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Evidence of metastatic disease.
* Patients will not require baseline staging PET or CT chest, abdomen, pelvis or bone scan to rule out metastatic disease prior to enrollment. Any staging scans will be ordered at the treating provider's discretion. If metastatic disease is found on any staging studies done, patients will not be eligible for enrollment.
* Locally advanced tumors at diagnosis (T4), including tumors fixed to the chest wall, peau d'orange, skin ulcerations/nodules, or clinical inflammatory changes (diffuse brawny cutaneous induration with an erysipeloid).
* Patients with stage III, HER2-negative cancer in the contralateral breast (see 3.1.6 above).
* Positive Hepatitis B (Hepatitis B surface antigen and antibody) and/or Hepatitis C (Hepatitis C antibody test) as indicated by serologies conducted ≤3 months prior to registration if liver function tests are outside of the normal institutional range.

NOTE: A hepatitis panel is required of all participants as part of screening. Patients with positive Hepatitis B or C serologies indicating active infection without known active disease must meet the eligibility requirements for ALT, AST, total bilirubin, INR, PTT, and alkaline phosphatase on at least two consecutive occasions, separated by at least 1 week. Patients with laboratory evidence of vaccination to Hepatitis B (e.g., positive antibodies) are eligible.

* Active liver disease, for example, due to autoimmune hepatic disorder, or sclerosing cholangitis.
* Significant, active cardiopulmonary dysfunction (i.e. uncontrolled heart issues)as indicated by MUGA or echocardiogram performed ≤60 days prior to registration and/or by presence of any of the following:

  * History of NCI CTCAE (Version 4.0) Grade ≥3 symptomatic congestive heart failure (CHF) or NYHA criteria Class ≥ II
  * Angina pectoris requiring anti-anginal medication, serious cardiac arrhythmia not controlled by adequate medication, severe conduction abnormality, or clinically significant valvular disease
  * High-risk uncontrolled arrhythmias (i.e., atrial tachycardia with a heart rate > 100/min at rest, significant ventricular arrhythmia [ventricular tachycardia], or higher-grade atrioventricular [AV]-block [second degree AV-block Type 2 [Mobitz 2] or third degree AV-block]); if adequately and safely treated, patient may be eligible.
  * Significant symptoms (Grade ≥ 2) relating to left ventricular dysfunction, cardiac arrhythmia, or cardiac ischemia
  * Myocardial infarction within 12 months prior to registration
  * Uncontrolled hypertension (systolic blood pressure > 180 mmHg and/or diastolic blood pressure >100 mmHg)
  * Evidence of transmural infarction on ECG
  * Requirement for oxygen therapy
* Co-morbid systemic illnesses or other severe concurrent disease which, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection or psychiatric illness/social situations that would limit compliance with study requirements.
* Currently receiving any other investigational agent which would be considered as a treatment for the primary neoplasm.
* Concurrent second malignancy or past malignancy with >30% estimated risk of relapse in next 5 years. EXCEPTIONS: Non-melanotic skin cancer or carcinoma-in-situ of the cervix in addition to smoldering pre-malignant or malignant conditions with minimized concern for clinical progression during treatment such as MGUS or CLL, based on treating provider's assessment. -NOTE: If there is a history or prior malignancy, patient must not be receiving active treatment for this malignancy cancer.
* Any prior treatment with T-DM1 or any trastuzumab therapy.
* Any neoadjuvant chemotherapy for this breast cancer.

  ->90 days of tamoxifen therapy, or other hormonal therapy, for adjuvant therapy for this malignancy
* NOTE: If the patient has received <90 days of such therapy but is still receiving it at the time of entry into the study, patient must temporarily stop the therapy prior to Cycle 1 Day 1. The therapy can re-start only after 6 weeks of T-DM1 have been administered (anytime after C3D1).
* History of exposure at any time to the following cumulative doses of anthracyclines:

  * Doxorubicin or liposomal doxorubicin >500mg/m2.
  * Epirubicin >900mg/m2.
  * Mitoxantrone >120 mg/m2.
  * Another anthracycline, or more than one anthracycline used in a cumulative dose exceeding the equivalent of doxorubicin 500mg/m2.
* History of intolerance (including Grade 3 or 4 infusion reactions) to murine proteins.
* History of previous invasive breast cancer ≤5 years.
* NOTE: History of DCIS, LCIS is allowed.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2018-08-22 (Actual); Primary Completion 2026-08-30 (Estimated); Study Completion 2029-08-30 (Estimated)

PRIMARY OUTCOMES:
5-year invasive disease-free survival rate | 5 years
  To evaluate invasive disease-free survival (IDFS) for patient receiving T-DM1

SECONDARY OUTCOMES:
Recurrence-free survival | 2 years
  To evaluate recurrence-free survival (RFS) for patient receiving T-DM1, defined as the time from study enrollment to disease recurrence and will not include death as an event.
Overall Survival | 2 years
  To evaluate overall survival (OS) for patient receiving T-DM1, defined as the time from study enrollment to death attributable to any cause (i.e. death from breast cancer, non-breast cancer cause, or from unknown cause).
Site of first recurrence | 2 years
  To evaluate site of first recurrence for patient receiving T-DM1, which will be tabulated as frequencies and relative frequencies.
Incidence Rate of each Toxicity (Safety) | 2 years
  To evaluate adverse events for patient receiving T-DM1, defined as adverse events of all grades utilizing CTCAE v4
Incidence Rate of Cardiac-Related Adverse Events (left ventricular systolic dysfunction) | 2 years
  To evaluate cardiac-related adverse events for patients receiving T-DM1, defined as incidence of symptomatic left ventricular systolic dysfunction
Incidence Rate of Cardiac-Related Adverse Events (cardiac death) | 2 years
  To evaluate cardiac-related adverse events for patients receiving T-DM1, defined as incidence of cardiac death
Incidence Rate of Cardiac-Related Adverse Events (decreased ejection fraction) | 2 years
  To evaluate cardiac-related adverse events for patients receiving T-DM1, defined as decrease in ejection fraction by at least 10 percentage points below baseline or to below 50%.

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Freedman, MD MPH, Principal Investigator — Dana-Farber Cancer Institute
Locations (14):
- United States (14):
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - The Stamford Hospital, Stamford, Connecticut
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute at St. Elizabeth's Medical Center, Brighton, Massachusetts
  - Dana-Farber/Brigham and Women's Cancer Center at Milford Regional Medical Center, Milford, Massachusetts
  - Dana-Farber/Brigham and Women's Cancer Center in clinical affiliation with South Shore Hospital, South Weymouth, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Dana-Farber/New Hampshire Oncology-Hematology, Londonderry, New Hampshire
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Rex Cancer Center, Raleigh, North Carolina
  - Lifespan Cancer Institute, Providence, Rhode Island
  - Sarah Cannon Research Institute, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No